CLINICAL TRIAL: NCT05975034
Title: Investigation of the Use of a Probiotic Supplement in People With Long COVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheffield Hallam University (Other)
Collaborators: Symprove UK (Unknown); Biomesight (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ER45883322
Record Dates: First submitted 2023-08-02; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Double-blinded randomised trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Computerised randomisation by a researcher in a separate department, probiotic/placebo packaged in identical bottles (label indicates group A or B). Probiotic/placebo delivered directly from supplier to participants (without involvement of the investigators).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Participants assigned to the probiotic group.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Participants assigned to the placebo group.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic taken daily for 12 weeks.
  Arms: Probiotic
Dietary Supplement: Placebo — Placebo taken daily for 12 weeks.
  Arms: Placebo

SUMMARY:
This study is a double-blinded randomised trial to assess the efficacy of a probiotic supplement in alleviating symptoms in people with Long COVID.

DETAILED DESCRIPTION:
240 participants with Long COVID will be randomly assigned to either a probiotic or placebo group in a 1:1 ratio for twelve weeks. Participants will track symptoms using an app for three weeks before the study, and for the last three weeks of the treatment. Participants will answer online questionnaires about their symptoms at 0, 4, 8, and 12 weeks. A subgroup of 60 participants will attend the laboratory for blood tests, cognitive function tests and gut microbiome analysis at 0 and 12 weeks. This group will also wear activity trackers for two weeks before the study, and for the final two weeks of the study.

ELIGIBILITY:
Inclusion Criteria: Long COVID defined as National Institute for Health and Care Excellence (NICE) criteria for Long COVID (Persistent symptoms at least 12 weeks after a confirmed or suspected Covid-19 infection).

-

Exclusion Criteria: Significant co-morbidities - no pre-existing diagnosis of hypertension, diabetes, cerebrovascular, cardiovascular or peripheral vascular disease, coagulopathy or haematological disorder or current or recent cancer.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-12-11 (Estimated); Study Completion 2023-12-11 (Estimated)

PRIMARY OUTCOMES:
Fatigue severity scale (FSS) | 12 weeks
  9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle
FACIT fatigue scale | 12 weeks
  Measure that assesses self-reported fatigue and its impact upon daily activities and function
EQ-5D-5L | 12 weeks
  Multi-attribute generic health status measure
Ability to Participate in Social Roles and Activities - PROMIS Short Form 8a | 12 weeks
  Evaluation of ability to participate in social roles and activities
Ecological Momentary Assessment (EMA) app | 12 weeks
  Symptom data collected using an app (sleep, fatigue, pain, breathlessness, light-headedness, cognitive difficulties)

SECONDARY OUTCOMES:
IBS-SSS | 12 weeks
  Composite score of abdominal pain, number of days with abdominal pain, bloating/distension, satisfaction with bowel habits, and IBS-related quality of life
Gastrointestinal Symptom Rating Scale | 12 weeks
  15 items in five symptom clusters: Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation
MRC Dyspnoea scale | 12 weeks
  Assesses the degree of functional disability due to dyspnoea
International. Physical Activity Questionnaire (short form) | 12 weeks
  Assesses moderate-to-vigorous physical activity and sedentary behaviour
Accelerometery data | 12 weeks
  Longitudinal measurement of movement
Cambridge Neuropsychological Test Automated Battery (CANTAB) | 12 weeks
  Computer-based cognitive assessment system
16S rRNA sequencing | 12 weeks
  Analysis of the composition and diversity of the gut microbiome
Analysis of inflammatory markers | 12 weeks
  Measurement of cytokines (including IL-8, IL-6) by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Dalton, PhD, Principal Investigator — Sheffield Hallam University
Locations (1):
- Sheffield Hallam University, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No